CLINICAL TRIAL: NCT04321759
Title: Comparative Effectiveness of Cognitive Enhancement Therapy vs. Social Skills Training in Serious Mental Illness
Brief Title: Comparative Effectiveness of CET vs. SST in SMI (Serious Mental Illness)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Matcheri S. Keshavan MD, Stanley Cobb Professor and Academic Head of Psychiatry, Department of Psychiatry,, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P000094; CER-2018C3-14701 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2020-03-18; First posted 2020-03-25 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Cognitive functioning; Social skills; Community functioning
MeSH Terms: conditions — Schizophrenia; Social Skills

STUDY DESIGN:
Intervention Model Description: Randomized cluster design with 19 service centers assigned to one of the two treatments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Enhancement Therapy (Experimental): CET is a comprehensive manualized cognitive remediation program designed to maximize gains in social functioning by integrating computer-based training to enhance neurocognition with group-based exercises to improve social cognition.
  Interventions: Behavioral: Cognitive Enhancement Therapy
- Social Skills Training (Active Comparator): The HOPES social rehabilitation program uses the principles of SST (modeling, role playing, positive and corrective feedback, homework assignments, in vivo skills practice), designed to improve both psychosocial functioning and preventive health..
  Interventions: Behavioral: Social Skills Training

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy — CET's group-based exercises are delivered for 1.5 hours each week in a group of 6-8 participants led by a clinician and an assistant, for one year. During each of three modules (basic concepts, social cognition, CET applications), the groups focus on acquisition of adult social milestones in perspective-taking, social context appraisal, and other aspects of social cognition, with psychoeducational lectures, homework assignments, and in-group exercises. Weekly supervision sessions for the clinician trainers will include review of how patients respond to the different demands of computer-based training and group-based exercises and guidance about improving engagement in both.
  Arms: Cognitive Enhancement Therapy
Behavioral: Social Skills Training — The psychosocial component involves weekly skills training classes delivered over one year, with modules including "Communicating Effectively," "Making and Keeping Friends," "Making the Most of Leisure Time," "Healthy Living," "Using Medications Effectively," and "Making the Most of a Health Care Visit" (Pratt et al., 2008). Participants attend two sessions each week (normally morning and afternoon of the same day): a 90-minute session focused on a specific skill and a 60-minute session in which the specific skill is used in role-play exercises.
  Other Names: HOPES
  Arms: Social Skills Training

SUMMARY:
To compare two evidence-based treatments, Cognitive Enhancement Therapy (CET) and Social Skills Training (SST) that have been shown in meta-analyses and in our own research to be effective to improve community functioning. The investigators will test the impact of CET and SST on community functioning, with special attention to their relative effectiveness for patients differing in baseline cognitive skills and age. The research uses a cluster design in which different mental health service centers are randomized to one of the two treatments.

DETAILED DESCRIPTION:
Aim 1. We will test our hypothesis that CET will be associated with greater improvements than SST in both the primary outcome: community functioning (SAS, QLS), and the secondary outcomes of neuro- and social cognition (NIH Toolbox, PennCNB, and MSCEIT) and social skills (SSPA). For study Aim 1, we hypothesized that CET will be associated with greater improvements than SST in both the primary outcome: community functioning (SAS, QLS), and the secondary outcomes of neuro- and social cognition (selected NIH Toolbox and Penn CNB measures, and MSCEIT) and social skills (SSPA). Aim 2: We will explore differential effectiveness of the two interventions by baseline cognitive functioning and age. For Aim 2, we hypothesize that patients with less impairment in cognitive functioning at baseline will demonstrate relatively larger treatment gains in SST compared to those in CET than those who are initially more cognitively impaired, and that younger patients will benefit more from CET compared to those in SST than those who are older. The results of this study will address a key knowledge gap in the field and a decisional dilemma for clinicians. A pilot study at four treatment sites will be used to test the feasibility and acceptability of telementalhealth delivery of these two treatments, as compared to in-person delivery.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 65;
2. DSM-5 diagnosis of schizophrenia or schizoaffective or schizophreniform disorder (confirmed via the MINI diagnostic interview);
3. estimated IQ of > 70 (established via WTAR).

Exclusion Criteria:

1. the presence of a current organic brain syndrome;
2. intellectual disability (DSM-5);
3. participation in either CET or SST within the prior year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Social Adjustment Scale II | Measurement at 0, 6, 12, 18, 24 months
  Measure of social functioning
Change in Heinrich Quality of Life Scale | Measurement at 0, 6, 12, 18, 24 months
  Measure of social functioning
Change in Social Skills Performance Assessment | Measurement at 0, 6, 12, 18, 24 months
  Measure of social functioning using role played scenarios

SECONDARY OUTCOMES:
Change in Auditory Verbal Learning Test | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of verbal ability in NIH Toolbox
Change in List Sorting Working Memory | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of working memory in NIH Toolbox
Change in Positive and Negative Syndrome Scale, PANSS-6 | Measurement at 0, 6, 12, 18, 24 months
  Short form of measure of positive and negative symptoms
Change in Picture Sequence Memory | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of visual/episodic memory & learning in NIH Toolbox
Change in Picture Vocabulary | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of language in NIH Toolbox
Change in Oral Reading Recognition | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of language in NIH Toolbox
Change in Penn Mouse Practice Test | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of speed of processing in PennCNB
Change in Penn Digit Symbol Test | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of speed of processing in PennCNB
Change in Penn Conditional Exclusion Test | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of reasoning & problem solving in PennCNB
Change in Penn Continuous Performance Test | Measurement at 0, 6, 12, 18, 24 months
  Neurocognition measure of reasoning & problem solving in PennCNB
Change in Managing Emotions | Measurement at 0, 6, 12, 18, 24 months
  Subscale of the Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT)

CONTACTS AND LOCATIONS:
Overall Officials: Matcheri S Keshavan, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Russell K Schutt, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - Hartford Hospital - Institute of Living, Hartford, Connecticut
  - Maine Medical Center, Portland, Maine
  - Massachusetts Mental Health Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schutt RK, Xie H, Mueser KT, Killam MA, Delman J, Eack SM, Mesholam-Gately R, Pratt SI, Sandoval L, Santos MM, Golden LR, Keshavan MS. Cognitive Enhancement Therapy vs social skills training in schizophrenia: a cluster randomized comparative effectiveness evaluation. BMC Psychiatry. 2022 Sep 1;22(1):583. doi: 10.1186/s12888-022-04149-x. PMID 36050663
- See also: Related Info — https://bmcpsychiatry.biomedcentral.com/counter/pdf/10.1186/s12888-022-04149-x.pdf